CLINICAL TRIAL: NCT05718713
Title: Respiratory Muscle Strength and Respiratory Functions in Patients With Chronic Low Back Pain
Brief Title: Respiration in Chronic Low Back Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seda Saka (Other)
Responsible Party: Sponsor-Investigator, Seda Saka, Asst. Prof., Halic University
Organization: Halic University (Other)
Other Study IDs: nterzikoparan1
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Chronic Low-back Pain
Keywords: Respiratory muscles; Respiratory function test; Muscle strength

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about respiratory muscle strength, respiratory functions, and balance in patients with chronic low back pain.

DETAILED DESCRIPTION:
Coordination between the stabilizer muscles of the trunk and respiratory functions may be lacking in people with chronic low back pain. However, a specially designed study investigating the relationship between respiratory functions and balance parameters in individuals with chronic low back pain is lacking. The goal of this observational study is to learn about respiratory muscle strength, respiratory functions, and balance in patients with chronic low back pain. Twenty-four individuals with low back pain for at least 6 months are going to include in the study. Pain assessment is going to assess with a Visual Analogue Scale. Respiratory muscle strength is going to measure by maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP). Pulmonary function assessment (PFT) is going to assess using a spirometer. Balance assessment is going to evaluate with Star Balance Test and Berg Balance Scale. Flexibility is going to evaluate with the Functional Reach Test.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with chronic low back pain
* being age 25-65
* defining pain with a minimum of 5 out of 10 in Visual Analog Scale (VAS)
* getting at least 24 points from the Mini Mental Test.

Exclusion Criteria:

* Having physical therapy in the last one month
* Orthopedic, neurological, and vestibular problems that will affect balance
* Severe discopathy
* Compression fracture
* Pregnancy
* Body Mass Index (BMI) of > 30kg

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic low back pain patients
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-04-20 (Estimated); Study Completion 2023-05-20 (Estimated)

PRIMARY OUTCOMES:
FEV1 (liter) | During the 6-month data collection process, pulmonary function measurements is going to made on the same day as the day the participants came to the clinic for examination or control.
  This is the amount of air with pulmonary function test that the patient can force out of their lungs in one second.
FEV1 (%-percentage) | During the 6-month data collection process, pulmonary function measurements is going to made on the same day as the day the participants came to the clinic for examination or control.
  This is the percentage of air with pulmonary function test that the patient can force out of their lungs in one second.
FVC (liter) | During the 6-month data collection process, pulmonary function measurements is going to made on the same day as the day the participants came to the clinic for examination or control.
  This is the greatest total amount of air patient can forcefully breathe out after breathing in as deeply as possible.
FVC (%-percentage) | During the 6-month data collection process, pulmonary function measurements is going to made on the same day as the day the participants came to the clinic for examination or control.
  This is the percentage of total amount of air patient can forcefully breathe out after breathing in as deeply as possible.
FEV1/FVC (percentage) | During the 6-month data collection process, pulmonary function measurements is going to made on the same day as the day the participants came to the clinic for examination or control.
  The FEV1/FVC ratio is a number that represents the percentage of patient lung capacity patient is able to exhale in one second.
Inspiratory muscle test | During the 6-month data collection process, pulmonary function measurements is going to made on the same day as the day the participants came to the clinic for examination or control.
  Maximal inspiratory pressure (MIP) is going to measured using a mouth pressure meter (MicroRPM; MicroMedical, UK) according to the guideline of ATS and European Respiratory Society (ERS).
Expiratory muscle test | During the 6-month data collection process, pulmonary function measurements is going to made on the same day as the day the participants came to the clinic for examination or control.
  Maximal expiratory pressure (MEP) is going to measured using a mouth pressure meter (MicroRPM; MicroMedical, UK) according to the guideline of ATS and European Respiratory Society (ERS).
Star Excursion Balance Test (SEBT) | During the 6-month data collection process, pulmonary function measurements is going to made on the same day as the day the participants came to the clinic for examination or control.
  Four strips of athletic tape will need to be cut to a length of 6-8 feet each. Two pieces will be used to form a '+', with the other two being placed over top to form an 'x' so that a star shape is formed. It is important that all lines are separated from each other by a 45° angle. The goal of the SEBT is to maintain single leg stance on one leg while reaching as far as possible with the contralateral leg.
  The person performing the test must maintain a their balance on one leg, while using the other leg to reach as far as possible in 8 different directions. The person (standing on his/her left leg for example) must reach in 8 different positions, once in each of the following directions: anterior, anteromedial, medial, posteromedial, posterior, posterolateral, lateral and anterolateral.
Berg Balance Scale (BBS) | During the 6-month data collection process, pulmonary function measurements is going to made on the same day as the day the participants came to the clinic for examination or control.
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete.

SECONDARY OUTCOMES:
Change in Visual Analog Scale (VAS) Pain Score | During the 6-month data collection process, pulmonary function measurements is going to made on the same day as the day the participants came to the clinic for examination or control.
  The VAS is a widely used scale for pain assessment in daily practice. VAS, with 0-10 numbers on it and they are asked to give a value between these numbers. 0: I have no pain, 10: I have very severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Seda Saka, Study Director; Abdullah Okur, Principal Investigator — XXX Clinic; Nagihan Koparan, Principal Investigator; Berna Calp, Principal Investigator
Locations (1):
- Haliç University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided